CLINICAL TRIAL: NCT03284034
Title: Comparison of the Efficacy Between Cryolipolysis Versus ATX-101 (Deoxycholic Acid) for the Treatment of Upper Back Fat: a Prospective Randomized Controlled Pilot Study.
Brief Title: Cryolipolysis Versus ATX-101 (Deoxycholic Acid) for Upper Back Fat
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll participants for analysis.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00205070
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Upper Back Fat
MeSH Terms: interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyrolipolysis (Active Comparator)
  Interventions: Device: CoolCurve
- Deoxycholic Acid (Experimental)
  Interventions: Drug: ATX-101

INTERVENTIONS:
Device: CoolCurve — The right and left sides of the upper back fat will be randomly assigned to receive Cryolypolysis (CoolCurve + Advantage applicator) 35 minutes session, 3 sessions 30 days apart.
  Other Names: CoolSculpt
  Arms: Cyrolipolysis
Drug: ATX-101 — The right and left sides of the upper back fat will be randomly assigned to receive The right and left sides of the upper back fat will be randomly assigned to receive ATX-101 (deoxycholic acid) injections, 3 sessions, 30 days apart.
  Other Names: Kybella
  Arms: Deoxycholic Acid

SUMMARY:
This is a prospective randomized controlled study comparing the efficacy of cryolipolysis versus ATX-101 (deoxycholic acid) for the treatment of upper back fat. Participants currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment. The treatment sites are the right and left upper back fat areas. The right and left sides of the upper back fat will be randomly assigned (1:1) to receive cryolipolysis, while the contralateral side will receive ATX-101.

This study was a pilot study designed to determine feasibility of this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years old
2. Subjects are in good health as judged by the investigator.
3. Subjects with mild to moderate upper back fat.
4. Subjects who are willing and have the ability to understand and provide informed consent for participation in the study and are able to communicate with the investigator.

Exclusion Criteria:

1. History of hypertrophic scars or keloids
2. Subjects currently under treatment with an antiplatelet or anticoagulant for any medical problem or patients who have coagulation disorder
3. Subjects who have a known history of cold-induced disease such as cryoglobulinemia, paroxysmal cold hemoglobulinuria, cold urticaria.
4. Pregnant or breast feeding
5. Uncooperative patients or patients with neurological disorders who are incapable of following directions or who are predictably unwilling to return for follow-up examinations.
6. Subjects who are unable to understand the protocol or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Change in fat measurements from baseline to Day 90. | Baseline and Day 90
  Subcutaneous fat measurement will be performed using an ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No